CLINICAL TRIAL: NCT06620484
Title: Musculoskeletal Ultrasound with Elastography in the Evaluation of Muscle State in Rheumatoid Arthritis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Kamel Khedr Mohamed, Resident, Assiut University
Other Study IDs: Musculoskeletal US in RA
Record Dates: First submitted 2024-08-06; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis; Musculoskeletal Ultrasound
Keywords: Muscle state
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis patients
  Interventions: Device: Musculoskeletal Ultrasound with elastography
- Healthy control group
  Interventions: Device: Musculoskeletal Ultrasound with elastography

INTERVENTIONS:
Device: Musculoskeletal Ultrasound with elastography — Musculoskeletal Ultrasound with elastography

SUMMARY:
Evaluation of muscle state in rheumatoid arthritis patients. Application of elastography in the detection of muscle stiffness in rheumatoid arthritis

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic debilitating disease. Muscle weakness is a common symptom in patients with rheumatoid arthritis (RA). From a metabolic perspective, muscle mass is determined by the balance between protein synthesis and degradation. People with RA note tenderness, stiffness, and pain in affected muscles.

In RA, chronic inflammation is a primary driver of muscle weakness. Persistent synovitis leads to the release of pro-inflammatory cytokines, such as tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6), which contribute to muscle atrophy and dysfunction. Joint damage and pain further limit physical activity, exacerbating muscle wasting through disuse atrophy. Additionally, the systemic inflammation associated with RA can lead to metabolic disturbances, including insulin resistance, which negatively impacts muscle protein synthesis and overall muscle health.

RA can cause a 25% to 70% reduction in muscular strength, typically caused by decreased skeletal muscle mass, ,Reduced muscle strength is usually considered to be a result of decreased muscle mass due to disuse atrophy. Rheumatoid cachexia, a term used in RA, is defined as a loss of skeletal muscle mass and with no, or little weight loss in fat mass Muscle weakness not only reduces the quality of life for the affected patients, but since patients' ability to work decreases it will also dramatically increase the burden on society (e.g. increased costs for long-term sick leave). Thus, RA severely affects both the individual and the society Given the complexity of muscle affection in RA , accurate assessment is essential for effective management. Conventional clinical methods, such as manual muscle testing and grip strength measurements, provide limited information on the underlying causes of muscle weakness. Advanced imaging techniques, such as conventional ultrasound (US) and shear wave elastography (SWE), offer a more comprehensive evaluation by providing detailed information on muscle morphology and stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18:70 years
* RA patients with positive RF And Anti ccp

Exclusion Criteria:

* History of injury or operation of the lower limb and upper limbs .
* History or clinical signs of neuromuscular disorders.
* Patients on drugs causing myopathy or myositis
* History of chronic diseases : kidney and liver disease
* Diabetic patients .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be divided into two groups matched for age and sex :
  Group A: rheumatoid arthritis will include 36 participants Group B: healthy participants (control) will include 36 participants
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of muscle state in rheumatoid arthritis patients by using musculoskeletal us | Baseline

SECONDARY OUTCOMES:
Application of elastography in the detection of muscle stiffness in rheumatoid arthritis patients | Baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frontera WR, Ochala J. Skeletal muscle: a brief review of structure and function. Calcif Tissue Int. 2015 Mar;96(3):183-95. doi: 10.1007/s00223-014-9915-y. Epub 2014 Oct 8. PMID 25294644
- [Background] Brennan FM, McInnes IB. Evidence that cytokines play a role in rheumatoid arthritis. J Clin Invest. 2008 Nov;118(11):3537-45. doi: 10.1172/JCI36389. PMID 18982160
- [Background] Huffman KM, Jessee R, Andonian B, Davis BN, Narowski R, Huebner JL, Kraus VB, McCracken J, Gilmore BF, Tune KN, Campbell M, Koves TR, Muoio DM, Hubal MJ, Kraus WE. Molecular alterations in skeletal muscle in rheumatoid arthritis are related to disease activity, physical inactivity, and disability. Arthritis Res Ther. 2017 Jan 23;19(1):12. doi: 10.1186/s13075-016-1215-7. PMID 28114971
- [Background] Londhe P, Guttridge DC. Inflammation induced loss of skeletal muscle. Bone. 2015 Nov;80:131-142. doi: 10.1016/j.bone.2015.03.015. PMID 26453502
- See also: Numbness, Muscle Pain, and Other RA Symptoms — https://www.healthline.com/health/symptoms-related-to-ra